CLINICAL TRIAL: NCT05332639
Title: Personalized Risk Estimation for Crohn's Disease (PRE-Crohn's): Implementation and Feasibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American College of Gastroenterology (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Emily R. Lopes, MD, MPH, Principal Investigator, Instructor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022p000905; 1K23DK136977-01 (NIH)
Record Dates: First submitted 2022-03-28; First posted 2022-04-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Crohn Colitis; Crohn's Ileocolitis; Crohn's Gastritis; Crohn's Jejunitis; Crohn's Duodenitis; Crohn's Esophagitis
Keywords: Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Personalized Risk Estimation for Crohn's Disease (PRE-Crohn's) tool
  Interventions: Behavioral: Personalized Risk Estimation for Crohn's Disease (PRE-Crohn's) tool
- Comparator arm (Active Comparator): Standard Crohn's Disease Education
  Interventions: Behavioral: Standard Crohn's Disease Education

INTERVENTIONS:
Behavioral: Personalized Risk Estimation for Crohn's Disease (PRE-Crohn's) tool — We will develop a web-based, personalized risk estimation for CD (PRE-Crohn's) tool to quantitate participants' relative risk (RR) and lifetime risk of CD based on known risk factors for disease. We will consider the following risk factors for Crohn's disease: body mass index (BMI); smoking history; NSAID use; intake of fruit, fiber, and added sugar; oral contraceptive use (females); antibiotic use; breast-feeding; pets in home; and anti-microbial biomarker positivity. This tool will also display a participants' personalized summary of their risk factors for CD as well as educational tools for modifying these factors. Construction of this tool is based on the Your Disease Risk tool developed by the Siteman Cancer Center at Washington University in St. Louis School of Medicine. The interventional group will also receive standard education about Crohn's disease (comparison group intervention) via the web-based tool.
  Other Names: Intervention Arm
  Arms: Intervention Arm
Behavioral: Standard Crohn's Disease Education — The comparison group will receive standard education about Crohn's disease, which will include information regarding the prevalence of disease, clinical presentation including signs and symptoms of disease, and treatment options including available medications. Upon completion of the study, the comparator arm will be given the option of receiving their personalized risk of Crohn's disease with the PRE-Crohn's tool as well.
  Other Names: Comparator Arm
  Arms: Comparator arm

SUMMARY:
The aim of this study is to develop and assess the feasibility and effect of a web-based, personalized risk-estimation for Crohn's disease (PRE-Crohn's) tool on behaviors and biomarkers associated with risk for Crohn's disease in unaffected first-degree relatives of patients with inflammatory bowel disease. We hypothesize that personalized risk disclosure via the PRE-Crohn's educational tool is both feasible and successful in modifying behaviors associated with Crohn's disease risk and normalizing pre-clinical disease biomarkers when compared to standard Crohn's disease education. Broadly, completion of this project will also help elucidate the role of lifestyle and dietary factors in pre-clinical Crohn's disease development in high-risk individuals, and provide novel insight into potential strategies for disease prevention in this population.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Ability and willingness to comply with all patient visits and study-related procedures
* Ability to understand and complete study questionnaires
* Must have at least one first-degree relative with inflammatory bowel disease (Crohn's disease, ulcerative colitis, or indeterminate colitis/IBD unclassified)
* Individuals greater than 14 years of age

Exclusion Criteria:

* Inability to provide informed consent
* Inability to comply with all patient visits and study-related procedures
* Inability to understand or complete study questionnaires
* Patients with existing diagnoses of inflammatory bowel disease (ulcerative colitis, Crohn's disease, or indeterminate colitis/IBD unclassified)
* Evidence of clinical signs or symptoms of inflammatory bowel disease, identified by a modified version of the Harvey-Bradshaw Index for CD activity

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Total enrollment (n) at 1.5 years and retention rate (%) at study conclusion | 1.5 years and time of study completion
  The total enrollment at 1.5 years and the retention rate recorded at the conclusion of the study will be measured based on completion of the 6-month survey.

SECONDARY OUTCOMES:
Motivation to change smoking behavior | 8 weeks and 6 months
  We will measure change in contemplation ladder scores for motivation to change smoking behavior (yes/no for achieving a 1-point increase)
Motivation to change diet | 8 weeks and 6 months
  We will measure change in contemplation ladder scores for motivation to change diet (yes/no for achieving a 1-point increase)
Motivation to change physical activity | 8 weeks and 6 months
  We will measure change in contemplation ladder scores for motivation to change physical activity (yes/no for achieving a 1-point increase)
Change in physical activity | 8 weeks and 6 months
  We will measure change in physical activity (MET-hours/week)
Change in fruit intake | 8 weeks and 6 months
  We will measure change in fruit intake (servings/day)
Change in vegetable intake | 8 weeks and 6 months
  We will measure change in vegetable intake (servings/day)
Change in processed meat intake | 8 weeks and 6 months
  We will measure change in processed meat intake (servings/day)
Change in fiber intake | 8 weeks and 6 months
  We will measure change in fiber intake (grams/day)
Change in added sugar intake | 8 weeks and 6 months
  We will measure change in added sugar intake (grams/day)
Change in smoking behaviors | 8 weeks and 6 months
  We will measure change in smoking behaviors including current smoking vs non-smoking and cigarettes/day
Change in C-reactive protein (CRP; mg/L) | 8 weeks and 6 months
  We will measure change in CRP (mg/L)
Change in fecal calprotectin (mcg/g) | 8 weeks and 6 months
  We will measure change in fecal calprotectin (mcg/g)
Change in seropositivity for antimicrobial biomarkers | 8 weeks and 6 months
  We will measure several Crohn's disease associated antimicrobial biomarkers including ASCA IgA and IgG, anti-OmpC, anti-CBir1, anti-A4-Fla2 and anti-FlaX will be assayed using the PROMETHEUS® IBD sgi Diagnostic® panel. Positivity for each of these components are defined as follows: ASCA IgA > 9.2 EU/mL; ASCA IgG > 11.9 EU/mL; anti-OmpC > 11.3 EU/mL; anti-CBir1 > 35.4 EU/mL; anti-A4-Fla2 > 32.4 EU/mL and anti-FlaX > 36.0 EU/mL. Total biomarker positivity (secondary outcome) will be defined as the presence of 1 or more positive individual biomarkers above. We will then assess for change in total biomarker positivity at 8 weeks and 6 months compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Lopes, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate-level results of from this study will be reported on clinicaltrials.gov. De-identified individual-level data will be uploaded to a separate controlled access repository and can be available upon reasonable request and per controlled access repository standard terms and procedures.
Time Frame: All scientific data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Access Criteria: A controlled repository will be used to store and protect individual patient data. To access data arising from this project, users must complete a data request form and Data Use Agreement (DUA), which limits subsequent use to the terms of the approved request and requires that users maintain data security, and refrain from any attempts to re-identify research participants or engage in any unauthorized uses of the data. To get access to the data, the user must submit a valid scientific question, include a statistical analysis plan.

REFERENCES:
- [Background] Colditz GA, Dart H. Commentary: 20 years online with "Your Disease Risk". Cancer Causes Control. 2021 Jan;32(1):5-11. doi: 10.1007/s10552-020-01356-3. Epub 2020 Oct 17. PMID 33068181
- See also: Your Disease Risk — https://siteman.wustl.edu/prevention/ydr/
- See also: NIH Reporter Prevention of Crohns Disease in High-Risk Individuals — https://reporter.nih.gov/search/EXri1pvFzUKQr3eynD7OnQ/project-details/10887042